CLINICAL TRIAL: NCT01875835
Title: Evaluation of Neointimal Coverage of Everolimus-Eluting Stent and Bare-metal Stent After Implantation in STEMI Patients by Optical Coherence Tomography
Brief Title: Evaluation of Neointimal Coverage of EES and BMS After Implantation in STEMI Patients by Optical Coherence Tomography
Acronym: NeoCover
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrolling the required number of participants has made it impractical to proceed with the trial.
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, The second affiliated hospitai of Harbin medical university, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMUOCT-STEMI
Record Dates: First submitted 2013-06-05; First posted 2013-06-12 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardiac infarction; Bare-metal stent; Everolimus-eluting stent; Optical coherence tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DES (Active Comparator): Everolimus-Eluting Stent implanted in patients with ST-segment elevation myocardial infarction (STEMI)
  Interventions: Device: Xience™ V stent (Abbott Vascular, Santa Clara, California, USA)
- BMS (Active Comparator): Bare-Metal Stent implanted in patients with ST-segment elevation myocardial infarction (STEMI)
  Interventions: Device: Multilink-Vision stent(Abbott Vascular, Santa Clara, California, USA)

INTERVENTIONS:
Device: Xience™ V stent (Abbott Vascular, Santa Clara, California, USA)
  Arms: DES
Device: Multilink-Vision stent(Abbott Vascular, Santa Clara, California, USA)
  Arms: BMS

SUMMARY:
Primary percutaneous coronary intervention (PCI) represents the preferred reperfusion strategy for patients with ST-segment elevation myocardial infarction (STEMI), since it is more effective than thrombolytic regimens in reducing adverse events, including death. Drug-eluting stents (DES) are currently being widely used in patients with STEMI. The effectiveness of DES to reduce restenosis and the need for revascularization compared with bare-metal stents (BMS) has been documented in randomized controlled trials. The first-generation DESs implanted in STEMI have been associated with delayed healing and incomplete strut coverage. Therefore, in patients with implanted DES, longer duration of dual antiplatelet therapy is needed. The second-generation DESs (ZES and EES) have been improved the drug and polymer, which have been proved to improve neointima healing compared with the first generation DESs.

However, the difference of strut coverage between EES and BMS implanted in STEMI patients is unknown. In this study, we assess the neointimal coverage at 3-month and 12-month follow-up in EES and BMS implanted in patients with STEMI by optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years
* Acute MI with ST-segment elevation, within 12 hours from symptoms onset.
* Length of culprit lesion≤25mm.
* Vessel size in between 2.5 and 4.0 mm.
* Signed patient informed consent.

Exclusion Criteria:

* Prior administration of thrombolytic therapy.
* Cardiogenic shock.
* Renal failure (Crea≥2.0mg/dL).
* Recent major bleeding.
* Allergy to heparin, aspirin, clopidogrel, everolimus, the polymer components of the Xience V stent, stainless steel, or contrast media.
* Left main disease
* Multi-vessel lesion
* Other hemodynamically significant lesion(s) is present in the infarct vessel (or side branches)
* Angiography demonstrates the infarct lesion to be at the site of a previously implanted stent or in bypass grafts.
* No suitable anatomy for OCT scan.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Comparison of the rate of covered struts to the EES vs BMS implanted in STEMI patients by frequency domain optical coherence tomography (FD-OCT). | 3-month
  The covered strut is defined as the strut has definite neointimal over it. And the rate of covered struts was calculated as the number of covered struts divided the number of total struts.

SECONDARY OUTCOMES:
Comparison of the rate of covered struts to the EES vs BMS implanted in STEMI patients by FD-OCT. | 12-month
  The covered strut is defined as the strut has definite neointimal over it. And the rate of covered struts was calculated as the number of covered struts divided the number of total struts.
Comparison of the rate of malaposed struts to EES vs BMS implanted in STEMI patients by FD-OCT. | 3-month
  Strut malapposition is defined as struts detached from the vessel wall > 108μm for EES and > 101μm for BMS. The rate of malaposed struts is calculated as the number of malaposed struts divided the number of total struts.
Comparison of the rate of malaposed struts to the EES vs BMS implanted in STEMI patients by FD-OCT. | 12-month
  Strut malapposition is defined as struts detached from the vessel wall > 108μm for EES and > 101μm for BMS. The rate of malaposed struts is calculated as the number of malaposed struts divided the number of total struts.
Major adverse cardiovascular events (MACE) | 12-month

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, MD,PhD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China